CLINICAL TRIAL: NCT01582763
Title: International GBS Outcome Study (IGOS): a Prospective INC Study on Clinical and Biological Predictors of Disease Course and Outcome in Guillain-Barré Syndrome (GBS).
Brief Title: International Guillain-Barré Syndrome Outcome Study
Acronym: IGOS
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B.C. Jacobs, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2011-477; 3290 (Other: Dutch Trial Registration)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Guillain-Barré Syndrome; Miller Fisher Syndrome
Keywords: Guillain-Barré syndrome; Polyneuropathy; Autoimmune Diseases; Immune System Diseases; Neuromuscular Diseases; Outcome; Quality of life; Disability; Prognostic Determinants; Treatment; Immunoglobulins; Prognosis; Infections; Anti-ganglioside antibodies; Genetic polymorphisms; Electrophysiology; Cerebrospinal Fluid; Serum
MeSH Terms: conditions — Guillain-Barre Syndrome; Miller Fisher Syndrome; Polyneuropathies; Autoimmune Diseases; Immune System Diseases; Neuromuscular Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, cerebrospinal fluid, samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- GBS: Guillain-Barré syndrome >1000, follow-up 1-3 years
- NC: Normal controls (NC)
- IC: Infectious controls (IC)
- OND: Other neurological diseases (OND)

SUMMARY:
International GBS Outcome Study (IGOS) is a study conducted by the members of the Inflammatory Neuropathy Consortium (INC) and Peripheral Nerve Society (PNS) on disease course and outcome in Guillain-Barré syndrome (GBS).

The IGOS aims to identify clinical and biological determinants and predictors of disease course and outcome in individual patients with Guillain-Barré syndrome, as early as possible after onset of disease.

DETAILED DESCRIPTION:
GBS is a post-infectious immune-mediated polyradiculoneuropathy with a highly diverse clinical course and outcome despite partially effective forms of treatment(immunoglobulins and plasma exchange). Outcome in patients with GBS has not improved in the last two decades. At present about 10 to 20% of patients remain severely disabled and about 5% die. One explanation for this stagnation is the highly variable clinical course of GBS and the lack of knowledge about the factors that determine the clinical course in individual patients with GBS. GBS may consist of distinct pathogenic subgroups, in which disease onset and progression is influenced by different types of preceding infections, anti-neural antibodies and genetic polymorphisms. Optimal treatment of individual patients may depend on the pathogenesis and clinical severity. Patients with severe forms of GBS may possibly need more intensive treatment to recover. Patients with a milder course that fully recover after standard therapy could suffer from possibly more side effects of more aggressive forms of treatment. This could only be possible if there are prognostic models that accurately predict the clinical course in individual patients. Ideally such models should be based on clinical and biological predictors that are strongly associated with disease course and known as early as possible in the acute phase of illness, when treatment with immunomodulatory therapy is most effective. Prognostic models could help to guide selective trials in specific GBS subtypes. Because of this it will be possible to treat GBS with more effective and more individual therapy.

This study aims to identify clinical and biological determinants and predictors of disease course and outcome in individual patients with Guillain-Barré syndrome, as early as possible after onset of disease. This information will be used to understand the diversity in clinical presentation and response to treatment of GBS. This information will also be used to develop new prognostic models to predict the clinical course and outcome accurately in individual patients with GBS.

To address these research questions it is required to conduct a prospective study with standardized collection of clinical data and biomaterials from a large group of well-defined GBS patients during a long follow-up period. Such an extensive study in a relatively rare disease as GBS can be addressed only by intensive international collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil diagnostic criteria for GBS of National Institute of Neurological Disorders and Stroke (NINDS). Patients with Miller Fisher syndrome and all other variants of GBS, including overlap syndromes, can be included.
* Inclusion of all males and females of all ages, independent of disease severity and treatment
* Inclusion within two weeks of onset of weakness
* Inclusion of patients transferred from another hospital if the stay in the first hospital was less than one week
* Opportunity to conduct a follow-up of at least one year
* Informed consent of patient or, in case of children, of parents or legal guardians

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Guillain-Barré syndrome (GBS) or variants of GBS, including the Miller Fisher syndrome (MFS) and overlap syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Guillain Barré Syndrome (GBS) disability score | 1 year
  7 scores for disability, ranging from a healthy state to dead; 0 = healthy state to 6 = dead
MRC sum score | 1 year
  the sum of MRC scores of six muscle groups, including shoulder abductors, elbow flexors, wrist extensors, hip flexors, knee extensors, and foot dorsiflexors on both sides, ranging from 60 (normal) to 0 (quadriplegic). 0 = no visible contraction to 5 = normal strength, score per muscle group

SECONDARY OUTCOMES:
Overall Neuropathy Limitations Scale (ONLS) | 1 year
  Questions regarding affection of ability in both arms and legs, with a score from 0 = normal to 5 = disability in both arms preventing all purposeful movements and a score from 0 = walking/climbing stairs/running not affected to 7 = restricted to wheelchair or bed most of the day, unable to make any purposeful movements of the legs
Fatigue Severity Scale (FSS) | 1 year
  the FSS is a simple and reliable instrument to assess and quantify fatigue for clinical and research purposes.
EurQol EQ-5D Health Questionnaire | 1 year
  EQ-5D® is a standardized instrument for use as a measure of health outcome with a scale from 0 = the worst health you can imagine to 100 = the best health you can imagine
Rasch-built Overall Disability Scale (R-ODS) | one year
  The R-ODS is a linearly weighted scale that specifically captures activity and social participation limitations in patients with GBS, CIDP, and MGUSP. Compared to the Overall Disability Sum Score, the R-ODS represents a wider range of item difficulties, thereby better targeting patients with different ability levels. If responsive, the R-ODS will be valuable for future clinical trials and follow-up studies in these conditions. Score from 0 = not possible to perform any activity to 48 = easy to perform any activity

CONTACTS AND LOCATIONS:
Overall Officials: Bart Jacobs, Dr., Principal Investigator — Erasmus Medical Center
Locations (138):
- United States (26):
  - Barrows Neurological Institute, Phoenix, Arizona
  - UC Irvine Health, Orange, California
  - Yale University School of medicine, New Haven, Connecticut
  - University of Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Lahey clinic Boston, Boston, Massachusetts
  - Tufts University School of Medicine, Boston, Massachusetts
  - Spectrum Health System, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - University at Buffalo, Buffalo, New York
  - Mt. Sinai School of Med, New York, New York
  - Columbia University, New York, New York
  - Montefiore MC, New York, New York
  - Wexner Medical Center at The Ohio State University, Columbus, Ohio
  - University of Tennessee, Memphis, Tennessee
  - UT Southwestern, Dallas, Texas
  - The university of Texas Health Science Center, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
- Argentina (7):
  - Hospital Austral, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Hospital Cesar Milstein, Buenos Aires
  - Hospital de Clinicas, Buenos Aires
  - Hospital Fleni, Buenos Aires
  - Hospital Garrahan, Buenos Aires
  - Hospital Militar, Buenos Aires
- Australia (2):
  - Royal Melbourne Hospital, Parkville, Victoria
  - Concord Repatriation General Hospital Sydney, Sydney
- Bangladesh (2):
  - Dhaka Medical College & Hospital, Dhaka
  - ICDDR,B, Dhaka
- Belgium (2):
  - Clinique Universitaire St. Luc, Brussels
  - University Hospital Leuven, Leuven
- Canada (4):
  - University of Calgary, Calgary
  - Queens University, Kingston
  - University hospital LHSC, London
  - University Health Network, Toronto
- China (4):
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiang Hospital Central South University, Changsha, Hunan
  - The affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
- Denmark (5):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - National Hospital Copenhagen, Copenhagen
  - Glostrup Hospital Copenhagen, Glostrup Municipality
  - Odense University Hospital, Odense
- France (4):
  - Hôpital St. Louis de Paris, Paris, Paris
  - Hospital de la Timone, Marseille
  - Nantes University Hospital, Nantes
  - University Strassbourg, Strasbourg
- Germany (6):
  - Universitätsklinikum der RWTH, Aachen
  - University of Cologne, Cologne
  - Universitatsklinikum Dresden, Dresden
  - Heinrich Heine University, Düsseldorf
  - University Hospital of Saarland, Homburg
  - Universitatsklinikum Würzburg, Würzburg
- University of Thessaly, Larissa, Thessaly, Greece
- Italy (11):
  - University of Genova, Genova
  - Ospedale Sant'Andrea La Spezia, La Spezia
  - Ospedale Luigi Sacco, Milan
  - Ospedale San Raffaele, Milan
  - University of Milan, Milan
  - University of Modena, Modena
  - University of Milano-Bicocca, Monza
  - Universita FedericoII di Napoli, Napoli
  - University of Padova, Padua
  - Policlinico Tor Vergata, Roma
  - Sant' Andrea Hospital, Rome
- Japan (6):
  - Chiba University School of Medicine, Chiba
  - Kinki University School of Medicine, Osaka
  - Hokkaido Medical Center, Sapporo
  - Dokkyo Medical Univeristy, Tochigi
  - National Defense Medical College, Tokorozawa
  - Toho University Medical Center, Tokyo
- University of Malaya, Kuala Lumpur, Malaysia
- Netherlands (19):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - AMC Amsterdam, Amsterdam
  - Gelre ziekenhuis, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Reinier de Graaf Groep, Delft
  - Van Weel-Bethesda Hospital, Dirksland
  - Albert Schweitzer Hospital, Dordrecht
  - Elkerliek hospital, Helmond
  - Westfriesgasthuis Hoorn, Hoorn
  - LUMC, Leiden
  - University Hospital Maastricht, Maastricht
  - CWZ Nijmegen, Nijmegen
  - Maasstad Hospital, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - SSVZ, Schiedam
  - HAGA ziekenhuis, The Hague
  - MCH Westeinde, The Hague
  - St. Elisabeth hospital, Tilburg
- University of Puerto Rico, San Juan, Puerto Rico
- University of Cape Town, Cape Town, South Africa
- Spain (10):
  - Hospital de Bellvitge, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Hospital 2 de Octubre, Madrid
  - Hospital Universitario Infanta Sofia, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Marques de Valdecilla, Santander
  - Hospital de Santiago, Santiago de Compostela
  - Hospital Virgen de Sevilla, Seville
- Switzerland (7):
  - Universityhospital Bern, Inselspital, Bern
  - HFR - Cantonal Hospital, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Lausanne University Hospital, Lausanne
  - Ospeale Civico Lugano, Lugano
  - Kantonspital St. Gallen, Sankt Gallen
  - Hopital du Valais, Sion
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (18):
  - Queen Elizabeth Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - University of Glasgow, Glasgow
  - Hinching Brooke Hospital, Huntingdon
  - NHS Forth Valley Hospital, Larbert
  - Leeds General Infirmary, Leeds
  - The Walton Centre, Liverpool
  - Charing Cross Hospital, London
  - King's College Hospital, London
  - National Hospital of Neurology and Neurosurgery, London
  - St. George's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle
  - University of Oxford, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doets AY, Lingsma HF, Walgaard C, Islam B, Papri N, Davidson A, Yamagishi Y, Kusunoki S, Dimachkie MM, Waheed W, Kolb N, Islam Z, Mohammad QD, Harbo T, Sindrup SH, Chavada G, Willison HJ, Casasnovas C, Bateman K, Miller JAL, van den Berg B, Verboon C, Roodbol J, Leonhard SE, Benedetti L, Kuwabara S, Van den Bergh P, Monges S, Marfia GA, Shahrizaila N, Galassi G, Pereon Y, Burmann J, Kuitwaard K, Kleyweg RP, Marchesoni C, Sedano Tous MJ, Querol L, Illa I, Wang Y, Nobile-Orazio E, Rinaldi S, Schenone A, Pardo J, Vermeij FH, Lehmann HC, Granit V, Cavaletti G, Gutierrez-Gutierrez G, Barroso FA, Visser LH, Katzberg HD, Dardiotis E, Attarian S, van der Kooi AJ, Eftimov F, Wirtz PW, Samijn JPA, Gilhuis HJ, Hadden RDM, Holt JKL, Sheikh KA, Karafiath S, Vytopil M, Antonini G, Feasby TE, Faber CG, Gijsbers CJ, Busby M, Roberts RC, Silvestri NJ, Fazio R, van Dijk GW, Garssen MPJ, Straathof CSM, Gorson KC, Jacobs BC; IGOS Consortium. Predicting Outcome in Guillain-Barre Syndrome: International Validation of the Modified Erasmus GBS Outcome Score. Neurology. 2022 Feb 1;98(5):e518-e532. doi: 10.1212/WNL.0000000000013139. Epub 2021 Dec 22. PMID 34937789
- [Derived] Jacobs BC, van den Berg B, Verboon C, Chavada G, Cornblath DR, Gorson KC, Harbo T, Hartung HP, Hughes RAC, Kusunoki S, van Doorn PA, Willison HJ; IGOS Consortium. International Guillain-Barre Syndrome Outcome Study: protocol of a prospective observational cohort study on clinical and biological predictors of disease course and outcome in Guillain-Barre syndrome. J Peripher Nerv Syst. 2017 Jun;22(2):68-76. doi: 10.1111/jns.12209. PMID 28406555
- See also: link to website — https://gbsstudies.erasmusmc.nl/